CLINICAL TRIAL: NCT06710990
Title: A Multicenter, Open-label, Fixed-sequence Study to Evaluate Drug-drug Interaction of Ritonavir and Itraconazole on the Pharmacokinetics of SHR-A1811 in Subjects With HER2-expressing Advanced Breast Cancer
Brief Title: Investigation of Drug-drug Interaction of Ritonavir and Itraconazole on the Pharmacokinetics of SHR-A1811 in Subjects With HER2-expressing Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-105
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Ritonavir; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: SHR-A1811 + Ritonavir (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Ritonavir
- Cohort 2: SHR-A1811 + Itraconazole (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Itraconazole

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811
Drug: Ritonavir — Ritonavir
  Arms: Cohort 1: SHR-A1811 + Ritonavir
Drug: Itraconazole — Itraconazole
  Arms: Cohort 2: SHR-A1811 + Itraconazole

SUMMARY:
The study is being conducted to evaluate the pharmacokinetics and safety of SHR-A1811 monotherapy and in combination with Ritonavir or Itraconazole in subjects with HER2-expressing advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score of 0 or 1;
2. Expected survival of not less than 3 months;
3. Important organ functions meet the following criteria:

   * Absolute neutrophil count (ANC) ≥1.5×109/L (1,500/mm3);
   * Platelet count (PLT) ≥100×109/L (100,000/mm3);
   * Hemoglobin (Hgb) ≥9.0 g/dL (90g/L);
   * Albumin level ≥3.0 g/dL;
   * Total serum bilirubin ≤1.5× the upper limit of normal (ULN);
   * Prothrombin time and activated partial thromboplastin time (aPTT) ≤1.5×ULN;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (for patients with liver metastasis, ALT and AST ≤5×ULN);
   * Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min;
   * QTcF ≤470 msec;
   * Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

1. Known active central nervous system metastases that have not been treated with surgery or radiation, except those that have been stable for at least 1 month after treatment and have discontinued corticosteroids for >2 weeks;
2. Having cardiac diseases, such as severe/unstable angina, symptomatic congestive heart failure (NYHA II-IV), clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, myocardial infarction within 6 months before the first administration, etc.
3. Known severe allergic history to any component of the SHR-A1811 product (ADC, total antibody, unconjugated toxin SHR169265 or its excipients), or hypersensitivity to humanized monoclonal antibody products (such as trastuzumab, pertuzumab, etc.);
4. Having contraindications to ritonavir or itraconazole use;
5. Having one or more factors that affect oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction, partial or total gastrectomy, etc.), or having active gastrointestinal diseases or other diseases that may significantly affect drug absorption, distribution, metabolism, or excretion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The maximum concentration (Cmax) for SHR-A1811 | Cycle 2 and Cycle 3. Each cycle is 21 days.
The maximum concentration (Cmax) for payload | Cycle 2 and Cycle 3. Each cycle is 21 days.
Area under the concentration curve from time 0 to 16 days (AUC0-16d) for SHR-A1811 | Cycle 2 and Cycle 3. Each cycle is 21 days.
Area under the concentration curve from time 0 to 16 days (AUC0-16d) for payload | Cycle 2 and Cycle 3. Each cycle is 21 days.

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | Cycle 2 and Cycle 3. Each cycle is 21 days.
Terminal half-life (t1/2) | Cycle 2 and Cycle 3. Each cycle is 21 days.
Area under the concentration curve from time 0 to infinity (AUCinf) | Cycle 2 and Cycle 3. Each cycle is 21 days.
Clearance (CL) | Cycle 2 and Cycle 3. Each cycle is 21 days.
Volume of distribution at steady state (Vss) | Cycle 2 and Cycle 3. Each cycle is 21 days.
Incidence and severity of adverse events | From the beginning of screening period to approximately 3 months after the last dose.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided